CLINICAL TRIAL: NCT07036471
Title: Evaluation of the myCare Start Service to Support Patients Starting a New Medicine in Switzerland: A Hybrid Type II Effectiveness-implementation Study
Brief Title: Supporting Patients Starting New Medicines: Evaluating the myCare Start Service in Switzerland
Acronym: myCare Start-I
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Geneva, Switzerland (Other)
Collaborators: University of Basel (Other); pharmaSuisse (Unknown); Center for Primary Care and Public Health (Unisante), University of Lausanne, Switzerland (Other); University of Bern (Other)
Responsible Party: Principal Investigator, Marie Paule Schneider, PhD, Prof. Dr. Marie Paule Schneider, University of Geneva, Switzerland
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Health Services Research
Other Study IDs: 2025-00715
Record Dates: First submitted 2025-05-12; First posted 2025-06-25 (Actual); Last update posted 2025-06-25 (Actual); Status verified 2025-04

CONDITIONS: Cardio-vascular Disease; Depression Disorders; Diabetes; COPD; Asthma Bronchiale; Hyperlipidaemia; Medication Initiation for Long-term Conditions
Keywords: patient adherence; medication adherence; medication initiation; long-term treatment; implementation science; interprofessional collaboration; outpatient care; community pharmacy; general practitioner; cost-effectiveness; medication adherence support programme
MeSH Terms: conditions — Diabetes Mellitus; Pulmonary Disease, Chronic Obstructive; Hyperlipidemias; Patient Compliance; Medication Adherence

STUDY DESIGN:
Intervention Model Description: Randomised stepped wedge cluster design study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual Care Arm (No Intervention): In the Usual Care Arm, the patients will receive the usual care from their pharmacist after being prescribed a new long-term medication.
- myCare Start Arm (Experimental): In the myCare Start Arm, the patients will receive the myCare Start service in their pharmacy after being prescribed a new long-term medication. myCare Start is an interprofessional health service offered by community pharmacies in Switzerland to support medication adherence in patients starting a new long-term treatment. It consists of two 10-minute, semi-structured and tailored consultations delivered by community pharmacists during the first 6 weeks of a patient initiating a new long-term medication, followed by tailored feedback to the patient's physician.
  Interventions: Behavioral: myCare Start

INTERVENTIONS:
Behavioral: myCare Start — The service consists of two 10-minute, semi-structured and tailored consultations delivered by community pharmacists during the first 6 weeks of a patient initiating a new long-term medication, followed by tailored feedback to the patient's physician.
  Arms: myCare Start Arm

SUMMARY:
In Phase B, the aim is to evaluate the myCare Start service in routine care within the ambulatory primary care medicine and community pharmacy setting in Switzerland. A Type II hybrid effectiveness-implementation study will be conducted to evaluate the effectiveness (improvement in adherence), cost-effectiveness and implementation of the service. This evaluation will allow us to build the necessary contextual relevant evidence base to support sustainable funding of the service in the long term.

DETAILED DESCRIPTION:
In Switzerland, almost half of the population has a long-term condition. Non-adherence to essential medication to treat these long-term conditions leads to suboptimal patient outcomes, increased hospitalisations, mortality, and financial burden to patients and healthcare systems. Innovative ways to address patient adherence within the ambulatory primary care medicine and community pharmacy setting in Switzerland are needed. Based on the UK New Medicine Service (NMS), pharmaSuisse introduced myCare Start into community pharmacy practice in Switzerland. However, like in other international settings barriers were experienced limiting its uptake and impact highlighting the need for context-based adaptation when the service is implemented in new settings. The myCare Start Implementation project (myCare Start-I) is a biphasic project to assist in optimising fit of the myCare Start service for Switzerland (Phase A) and evaluate its impact (Phase B). In Phase A, which is now complete, using implementation science methods, researchers conducted a thorough contextual analysis of the Swiss primary care ecosystem and adapted the existing myCare Start model using an iterative co-creation process with stakeholders to suit the needs of the primary care context. In Phase B a Type II hybrid effectiveness-implementation study will be conducted to evaluate the effectiveness (improvement in adherence), cost-effectiveness and implementation of the service to build the necessary evidence base to support sustainable funding of the service in the long term.

ELIGIBILITY:
Patients

Inclusion Criteria:

* Must have mandatory basic health insurance in Switzerland
* Must have been newly prescribed one or more new long-term medications in accordance with the following chronic conditions: cadisovascular diseases (incl. hyertension and thromboprophylaxis), diabetes, hyperlipidemia, depression, respiratory illness (asthma and COPD)
* Must be able to self-manage treatment (i.e. they live at home without any support to manage their medication, exception: patient uses a pill dispenser and fills it in by him-/herself)
* Must be able to understand language spoken by pharmacy staff and can read and understand study documents (French, German, English)
* Must understand and are willing to consent to the myCare Start-I study (including the agreement on self-reported questionnaires and collection of health care data via their health insurance company)
* in the intervention arm, patients must receive the myCare Start service

For this study, a new medication is a medication that has not been previously dispensed to the patient. This includes one or more new medications for a new diagnosis and or new medications for pre-existing diagnosis of a long-term condition. Included in this working definition:

* The new medication is indicated for one of the five long-term diseases listed above
* Patient has never had this active ingredient dispensed before (patient still considered eligible if they have received a small initial sample pack from their physician) or restarts an active ingredient after a period of interruption of at least 12 months (time period to be reported by the patient). Please note that for patients, that have already started a sample pack of medication the myCare Start Consultation One can start upon first dispensation at the pharmacy, there is no need to wait 7-14 days.
* The new active ingredient can be part of a combo preparation (e.g. a diuretic added to an ACE inhibitor into the same preparation)
* Patient has had no change in active ingredient but has an important change in treatment administration, such as:

  * Change of galenic form (e.g. two different types of inhalators for asthma/COPD)
  * Intensification of dosage regiment (e.g. twice a day instead of once a day)
* The following change is not considered as medication initiation:

  * New dosage of already known active ingredient (e.g. dose escalation of antidepressants)
  * Simplification of administration mode (e.g. metformin 1000 mg 1-0-0 instead of 500 mg 1-0-1; change in antihypertensive drug regiment in elderly patients having vertigo in the morning: 0-0-X instead of X-0-0)

Exclusion Criteria:

* Patients participating or having participated in an education program about their disease or treatment in the last 3 months, led by healthcare providers such as physicians, nurses, pharmacists or other (e.g. education provided by nurses for type I diabetes patients)

Physicians:

Inclusion criteria

- Any physician treating a patient for one of the five long-term illnesses listed above is eligible to refer the patient to a pharmacy providing myCare start.

Pharmacies:

Inclusion criteria:

* Have to be enrolled into the myCare Start service and comply to the requirements of the pharmacy quality system management of having access to a private consultation room or area
* Must agree to participate in the research study, including the recruitment of control patients and the delivery of the myCare Start service to intervention patients.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1600 (Estimated)
Dates: Start 2025-06 (Estimated); Primary Completion 2027-01 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Medication adherence (subjective measure) | Surveys at 14 days, 6 weeks, 3, 6 and12 months upon enrollement.
  Patient self-reported (subjective measure): We will use the BAASIS© (Basel Assessment of Adherence to Immunosuppressive Medications Scale), a 6-item scale with demonstrated psychometric properties in transplantation and other chronic diseases, as it assesses adherence according to the ABC taxonomy (Initiation, Medication Implementation, and Persistence). The BAASIS scale has a minimum and maximum value of 6 and 30, respectively. Lower scores on the BAASIS indicate poorer adherence to immunosuppressive medications, while higher scores indicate better adherence. This self-report instrument consists of six items that assess different aspects of medication adherence, including dose taking, drug holidays, timing deviation, reduction of dose, persistence, and timing of dose taking.

SECONDARY OUTCOMES:
Medication adherence (objective measure) | Form 1 month prior to enrollement up to 12 months after enrollment of the patient in the study.
  Prescription renewal records (objective measure): Medication renewal records will be extracted from health insurance data and analyzed using the "AdhereR" software in R.
Cost-effectiveness short-term | 12 months upon enrollment
  Total healthcare utilisation, in terms of total costs per patient, will be evaluated over the duration of the myCare Start follow-up period (12 months) using health insurance data. This will be combined with adherence results to determine the incremental cost-effectiveness ratio between the total costs per patient in the intervention vs. the control groups and the difference in adherence between groups. The survey will be forwarded to the patient at 14 days, 6 months, and 12 months after inclusion into the study via an emailed online survey. The main analysis consists of calculating 1) the incremental cost-effectiveness ratio between the total costs per patient in the intervention vs. the control group and 2.) the difference in adherence between groups and the probability that the intervention is cost-effective when the willingness to pay varies (i.e. the cost-effectiveness acceptability curve), the two classic indicators of cost-effectiveness analyses of health programmes.
Cost-effectiveness long-term | Calculations will be conducted during the 12-month follow-up phase
  Long-term potential healthcare cost savings will be evaluated using Markov Modelling. The Markov Modelling approach applied in this study is an adapted version of the models previously used in the UK to evaluate the New Medicine Service, adjusted with parameters tailored to the Swiss context. This approach will enable the projection and estimation of medium- and long-term benefits arising from improved adherence to the prescriptions as a result of the myCare start intervention. In Switzerland, the most commonly prescribed medications for long-term illnesses include cholesterol-lowering therapies, type 2 diabetes drugs, hypertension treatments, and antidepressants. For these four medication groups, specific Markov models have been developed. These calculations will be conducted during the 12-month longitudinal follow-up phase.
Implementation Outcome: Acceptability | - Every 2 months during the intervention phase of the study (for pharmacies and physicians) - at 2 & 6 weeks, 3, 6 and 12 months upon inclusion for intervention patient.
  The AIM (=Acceptability of Intervention Measure) will be used.
Implementation Outcome: Appropriateness | - Every 2 months during the intervention phase of the study (for pharmacies and physicians) - at 2 & 6 weeks, 3, 6 and 12 months upon inclusion for intervention patient.
  The IAM (=Intervention Appropriateness Measure) will be used.
Implementation Outcome: Feasibility | - Every 2 months during the intervention phase of the study (for pharmacies and physicians) - at 2 & 6 weeks, 3, 6 and 12 months upon inclusion for intervention patient.
  The FIM (=Feasibility of Intervention Measure) will be used.
Implementation Outcomes: Implementation cost | Throughout the duration of the study - approximately 12 months
  Cost of implementation will be assessed using the time-driven activity-based cost (TDABC) instrument. This pragmatic method allows investigators to systematically estimate the cost of implementation strategies (e.g. training, reorganisation of practice, regular stakeholder meetings) and the cost of the intervention.
Implementation Outcomes: Adoption | Throughout the duration of the study - approximately 12 months
  Adoption is defined as "the intention, initial decision, or action to try or employ an innovation or evidence-based practice".
  It will be measured through investigator onboarding logs and consultation records (No. of invited pharmacies and physicians, No. who completed training, No. who recruited or referred patients, No. of patients who participated in the intervention).
Implementation Outcomes: Fidelity | During the intervention phase of the pharmacies - approximately 12 months
  Fidelity is defined as the degree to which an intervention was implemented as it was prescribed in the original protocol.
  Consultation records (from the myCare Start consultations) and facilitation checklists will be used, to understand if the service is being carried out as intended and in appropriate areas.

CONTACTS AND LOCATIONS:
Overall Officials: Marie Paule Schneider, Prof. PhD, Principal Investigator — Uinversity of Geneva
Locations (1):
- Université de Genève, Geneva, Canton of Geneva, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided
Once fully anonymized, quantitative data will be annotated and structured to make them sharable, and registered in a FAIR-compliant data repository.